CLINICAL TRIAL: NCT03804619
Title: Accelerated Intermittent Theta-Burst Stimulation for Opiate Use Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled. No longer continuing study.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Gregory Sahlem, Assistant Professor, Department of Psychiatry and Behavioral Sciences, Stanford University, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 48431
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Opiate Dependence; Suicidal Ideation; Depression; Opioid Use; Opioid-Related Disorders; Opioid-use Disorder; Major Depressive Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Suicidal Ideation; Depression; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Open label, two-site randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Left DLPFC aiTBS stimulation (Experimental): Participants will receive aiTBS (intermittent theta burst stimulation) to a brain area called the left dorsolateral prefrontal cortex (L-DLPFC). Stimulation intensity will be individualized according to the individual's resting motor threshold.
  Interventions: Device: Accelerated intermittent theta-burst stimulation (aiTBS)
- ACC aiTBS stimulation (Experimental): Participants will receive aiTBS (intermittent theta burst stimulation) to a brain area called the anterior cingulate cortex (ACC). Stimulation intensity will be individualized according to the individual's resting motor threshold.
  Interventions: Device: Accelerated intermittent theta-burst stimulation (aiTBS)

INTERVENTIONS:
Device: Accelerated intermittent theta-burst stimulation (aiTBS) — aiTBS is an effective form of non-invasive brain stimulation which has been FDA-approved for the treatment of Major Depressive Disorder (MDD)

SUMMARY:
This study aims to examine whether multiple spaced sessions of intermittent theta-burst transcranial magnetic stimulation (iTBS) induce anti-depressant responses and reduce opiate cravings in adults with opiate use disorder (OUD). Additionally, we hope to identify whether the effectiveness of iTBS is related to changes in functional connectivity between particular brain areas.

DETAILED DESCRIPTION:
The proposed study aims to investigate the effectiveness of aiTBS applied to either the L-DLPFC or the ACC for reducing SI in individuals with OUD and identify neural functional connectivity changes underlying treatment response. 30 individuals with OUD who endorse suicidal ideation will be recruited. The accelerated iTBS treatment will involve 10 daily sessions of iTBS. Stimulation will be delivered to either the ACC or the L-DLPFC for 5 consecutive days. Suicidal ideation, depressive symptoms and opiate misuse will be measured before and after the 5-day stimulation course. Functional magnetic resonance imaging (fMRI) scans will also be carried out before and after stimulation to examine aiTBS-induced changes in neural functional connectivity. Changes in suicidal ideation, depressive symptoms and opiate misuse will be measured using both clinician-rated and self-report assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 at the time of screening
2. Able to read, understand, and provide written, dated informed consent prior to screening. Participants will be deemed likely to comply with study protocol and communicate with study personnel about adverse events and other clinically important information.
3. Diagnosed with Opiate Use Disorder, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders.
4. Endorse suicidal ideation (score >2 on the SSI-C).
5. Not in a current state of mania or psychosis (Young Mania Rating Scale)
6. In good general health, as ascertained by medical history.
7. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following specific criteria:, a. Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized (status post hysterectomy, bilateral tubal ligation), or is post-menopausal with her last menses at least one year prior to screening); or, b. Childbearing potential, and meets the following criteria. Childbearing potential, including women using any form of hormonal birth control, on hormone replacement therapy started prior to 12 months of amenorrhea, using an intrauterine device (IUD), having a monogamous relationship with a partner who has had a vasectomy, or is sexually abstinent. ii. Negative urinary pregnancy test at screening, confirmed by a negative urinary pregnancy test at randomization prior to receiving study treatment. iii. Willing and able to continuously use one of the following methods of birth control during the course of the study, defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly: implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence. The form of birth control will be documented at screening and baseline.
8. Clear urine drugs test
9. Registered with a psychiatrist
10. On stable psychotropic medication or psychotherapy for at least 6 weeks prior to the study with plans to continue throughout study enrollment.
11. Failed at least one anti-depressant trial (>/=6 week duration at an effective dose)
12. Ability to tolerate clinical study procedures.
13. No contraindications for TMS or MRI

Exclusion Criteria:

1. Any abnormalities indicated on the MRI e.g. structural neurological condition, more subcortical lesions than would be expected for age, stroke effecting stimulated area or connected areas or any other clinically significant abnormality that might affect safety, study participation, or confound interpretation of study results.
2. Metal implant in brain (e.g. deep brain stimulation), cardiac pacemaker, or cochlear
3. History of epilepsy/ seizures (including history of withdrawal/ provoked seizures)
4. Shrapnel or any ferromagnetic item in the head.
5. Pregnancy
6. Autism Spectrum disorder
7. Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
8. Active substance use (<1 week) or intoxication verified by toxicology screen--of cocaine, amphetamines, benzodiazepines
9. Cognitive impairment (including dementia)
10. Current severe insomnia (must sleep a minimum of 5 hours the night before stimulation)
11. Current mania
12. Current unmanageable psychosis
13. Showing symptoms of withdrawal from alcohol or benzodiazepines
14. IQ<70
15. Movement disorder
16. Any other indication the PI feels would comprise data.
17. Motor threshold value which does not enable treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Change in Beck Scale for Suicidal Ideation (SSI) score | After all stimulation sessions have been completed (approximately 48 hours after the final session)
  19-item clinician administered assessment to measure the intensity, pervasiveness, and characteristics of suicidal ideation in adults. Scores range from 0-38.

SECONDARY OUTCOMES:
Change in Columbia Suicide Severity Scale (C-SSRS) score | After all stimulation sessions have been completed (approximately 48 hours after the final session)
  Self-report measure for suicidal ideation
Change in Obsessive compulsive drug-use scale (OCDUS) score | After all stimulation sessions have been completed (approximately 48 hours after the final session)
  Self-report measure of drug craving. This questionnaire will be adapted to make it specific for opiate use.
Change in Montgomery Asberg Depression Rating Scale (MADRS) score | After all stimulation sessions have been completed (approximately 48 hours after the final session)
  A 10-item clinician-administered scale, designed to be particularly sensitive to antidepressant treatment effects in patients with major depression. Severity gradations for the MADRS have been proposed: 9-17 = mild depression, 18-34 = moderate depression, and ≥ 35 = severe depression. Scores range from 0-60.
Change in Beck Depression Inventory II (BDI-II) score | After all stimulation sessions have been completed (approximately 48 hours after the final session)
  The Beck Depression Inventory (BDI-II) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. BDI-II items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63.
Change in resting-state functional connectivity. | After all stimulation sessions have been completed (approximately 48 hours after the final session)
  Resting-state fMRI scans will be conducted before and after the course of aiTBS to examine changes in resting-state functional connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sahlem, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No